CLINICAL TRIAL: NCT01705002
Title: A Phase I, Dose-Escalating, Safety Study of an Intravenously Administered Pegylated Liposomal Mitomycin-C Lipid-based Prodrug (PL-MLP, PROMITIL) in Cancer Patients With Solid Tumors.
Brief Title: Intravenously Administered Pegylated Liposomal Mitomycin-C Lipid-based Prodrug (PROMITIL) in Cancer Patients With Solid Tumors.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lipomedix Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROMITIL-01
Record Dates: First submitted 2012-10-08; First posted 2012-10-12 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Cancer; Solid Tumor; Metastatic Colorectal Cancer (mCRC)
Keywords: phase 1; dose escalating; prodrug; mitomycin C; Capecitabine
MeSH Terms: conditions — Neoplasms; Colorectal Neoplasms | interventions — Capecitabine; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (12):
- Cohort A: Promitil 0.5 mg/kg (Experimental): Three treatment cycles, intravenous infusion of Promitil
  Interventions: Drug: Promitil
- Cohort B: Promitil 1.0 mg/kg (Experimental): Three treatment cycles, intravenous infusion of Promitil
  Interventions: Drug: Promitil
- Cohort C: Promitil 1.5 mg/kg (Experimental): Three treatment cycles, intravenous infusion of Promitil
  Interventions: Drug: Promitil
- Cohort D: Promitil 2.0 mg/kg (Experimental): Three treatment cycles, intravenous infusion of Promitil
  Interventions: Drug: Promitil
- Cohort E: Promitil 2.5 mg/kg (Experimental): Three treatment cycles, intravenous infusion of Promitil
  Interventions: Drug: Promitil
- Cohort F: Promitil 3.0 mg/kg (Experimental): Three treatment cycles, intravenous infusion of Promitil
  Interventions: Drug: Promitil
- Cohort G: Promitil 3.5 mg/kg (Experimental): Three treatment cycles, intravenous infusion of Promitil
  Interventions: Drug: Promitil
- Cohort H: Promitil 4.0 mg/kg (Experimental): Three treatment cycles, intravenous infusion of Promitil
  Interventions: Drug: Promitil
- Expanded Cohort (Experimental): Patients treated with the selected RP2D of PROMITIL (3 mg/kg) intravenously administered on their first cycle and reduced dose of 2 mg/kg from cycle 2 and onwards.
  Only for mCRC patients.
  Interventions: Drug: Promitil
- Combination Cohort (Experimental): Patients treated with one cycle of 2.5mg/kg Promitil day 1 together with Capecitabine 1,000 mg bid po days 1-21 followed by two cycles of 2.0 mg/kg Promitil day 1 together with Capecitabine 1,000 mg bid po days 1-21, at four-week intervals.
  Only for mCRC patients.
  Interventions: Drug: Promitil; Drug: Capecitabine
- Triple combination Cohort (Experimental): Patients treated with one cycle of 2mg/kg Promitil I.v and 5 mg/kg Bevacizumab i.v on day 1 together with Capecitabine 1,000 mg bid p.o days 1-14 at four-week intervals.
  Only for mCRC patients.
  Interventions: Drug: Promitil; Drug: Capecitabine; Drug: Bevacizumab
- 3 Weekly Cohort (Experimental): Patients treated with one cycle of 2mg/kg Promitil I.v and 7.5 mg/kg Bevacizumab i.v on day 1 together at three-week intervals.
  Only for mCRC patients.
  Interventions: Drug: Promitil; Drug: Bevacizumab

INTERVENTIONS:
Drug: Promitil — 2 mg/kg dose IV
Drug: Capecitabine — 1000 mg dose BID PO for days 1-21 for Combination Cohort and on day 1-14 on Triple combination Cohort
  Other Names: Xeloda
  Arms: Combination Cohort; Triple combination Cohort
Drug: Bevacizumab — for Triple combination cohort an IV dose of 5 mg/kg on day 1 at 4 week interval. For the 3 weekly cohort an IV dose of 7.5 mg/kg at 3 week interval.
  Other Names: Avastin
  Arms: 3 Weekly Cohort; Triple combination Cohort

SUMMARY:
This is a Phase I, multi-center, Dose-Escalating, Safety Study of an Intravenously Administered Pegylated Liposomal Mitomycin-C Lipid-based Prodrug (PL-MLP, PROMITIL) in Cancer Patients with Solid Tumors. The study comprised of:

Escalated cohorts A-H: 27 male or female participants, ages 18-80, BMI 18-36 diagnosed with inoperable, recurrent or metastatic malignant solid tumors, deemed incurable, and who have failed to respond to standard therapy or for whom no standard therapy is available. Eligible subjects will be assigned, successively in order of accrual, to one of eight cohorts, to receive escalating doses of intravenously infused PROMITIL. PROMITIL will be administered as an intravenous infusion. Dose escalation will only proceed in the absence of dose-limiting toxicity (DLT). For this purpose, each cohort will only begin its first cycle of PROMITIL when the cohort preceding it has successfully completed its first 4-week cycle without any signs of DLT.

Expanded cohort: 17 adult patients with metastatic CRC. The purpose of this expanded cohort is to further evaluate the safety of Promitil and to search for signs of antitumor activity of Promitil in this specific patient population.

Combination Cohort (Promitil concomitantly with Capecitabine): 23 adult patients with metastatic CRC.

Triple combination Cohort: 13 additional subjects with metastatic CRC, received combination of Promitil concomitantly with Bevacizumab (5 mg/kg) on day 1 of a 28 day cycle and Capecitabine on days 1-14 of a 28 day cycle.

3 weekly cohort- 9 subjects with metastatic CRC will receive Promitil and Bevacizumab (7.5 mg/kg) on day 1 of a 21 day cycle.

DETAILED DESCRIPTION:
For all cohorts, PROMITIL will be administered as an intravenous infusion at an initial rate of 0.25mg/min followed by gradual increase to a maximal rate of 2mg/min until completion of dosing, if absence of infusion reactions is established and in line with most updated version of IFU available for this study.

For each subject, subsequent dosing will take place 28 days after the previous treatment, provided they are deemed fit to be dosed again.

Patients will return to the study center on days 8, 15, 22 of cycle 1, and on day 15 of cycles 2 and 3, for monitoring assessments.

All patients will be followed-up for survival and post-Promitil treatment. Patients who did not received 3 cycles of PROMITIL will be followed up only until PD.

For the 3 weekly cohort Promitil will be administered at 3 week interval together with Bevacizumab (7.5 mg/kg). Patients will return to the study center on days 8 and 15 of cycle 1, and on day 15 of cycles 2 and 3, for monitoring assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with inoperable, recurrent or metastatic malignant solid tumors, deemed incurable, and who have either:

   * Failed to respond to standard therapy or
   * For whom no standard therapy is available or
   * Refuse to receive standard therapies
2. Histologically or cytologically confirmed diagnosis of solid tumor on file.
3. Age 18-80 years
4. BMI: 18-36
5. ECOG Performance Status ≤ 2
6. Estimated life expectancy of at least 3 months
7. Adequate bone marrow function (an absolute neutrophil count ≥1500/mm3, hemoglobin ≥9.5 g/dl, HgbA1C≤7%, and a platelet count ≥100,000/mm3(
8. Adequate liver function (serum bilirubin ≤2.0 mg/100 ml; alanine aminotransferase ≤2× ULN)
9. Adequate renal function (serum creatinine ≤1.5 mg/100 ml or creatinine clearance ≥45 ml/min/1.73m2)
10. No prior intravenous treatment with Mitomycin-C either alone or in combination
11. No other myelosuppressive treatment within 4 weeks before start of the study drug.
12. No other anti-cancer treatment within 2 weeks before start of the study drug
13. No prior extensive radiotherapy (e.g., whole pelvis total neuroaxis or greater than 50% of neuroaxis, whole abdomen, whole body or half-body) or bone marrow transplantation with high dose chemotherapy and/or total body irradiation. Re-irradiation of a field in abdomen/pelvis will be considered as extensive radiotherapy, excluding such patients from the study.
14. Women of child bearing potential practicing an acceptable method of birth control.
15. Understanding of study procedures and willingness to comply for the entire length of the study and to give written informed consent.
16. Additional criteria only for the Expanded Cohort and both Combination cohorts: Patients with histologically or cytologically confirmed recurrent and/or metastatic measurable or nonmeasurable CRC, with tissue or cytological diagnosis of cancer on file.
17. Additional criteria only for the Expanded Cohort and both Combination cohort: Patients who demonstrated either progression or intolerance when treated with irinotecan and fluopyrimidine-based chemotherapy, and, in the case of K-ras wild type tumors, anti-EGFR antibodies (Cetuximab, Panitumumab). Prior treatment with oxaliplatin or bevacizumab is allowed but not required.
18. Additional criteria only for the Expanded Cohort and both Combination cohorts: A ≥28 day treatment-free interval between last chemotherapeutic treatment and first treatment with Promitil, with the exception of Capecitabine and biological therapies, where 14-day treatment-free intervals suffice. this is also relevant for patients in the Combination Cohort that are currently taking Capecitabine prior to enter the study).
19. Additional criteria for the Triple Combination Cohort with bevacizumab only: Prior exposure to oxaliplatin should have terminated at least 6 months before start of PROMITIL, whether given as adjuvant therapy or as therapy for metastatic disease.
20. Additional criteria for the triple Combination Cohort with bevacizumab only: A ≥ 28 day treatment-free interval from last bevacizumab treatment

Exclusion Criteria:

1. Known hypersensitivity to the study drug or to any of its components
2. CHF (NYHA = Class IV) or LVEF≤40%
3. COPD > Stage 3 (FEV1<50%, FEV1/FVC<70%);
4. Cirrhosis (Child-Pugh Class C score);
5. Serum Albumin level < 3 g/dl
6. Any other severe concurrent disease which in the judgment of the investigator would make the subject inappropriate for entry into this study
7. History of human immunodeficiency virus (HIV) infection
8. History of chronic active hepatitis including subjects who are carriers of hepatitis B virus (HBV) or hepatitis C virus (HCV).
9. Presence of uncontrolled infection.
10. Evidence of active bleeding or bleeding diathesis
11. Brain metastases in symptomatic patients requiring ≥4 mg dexamethasone/day. However, patients with treated brain metastases by surgery or radiation who are stable and symptom-free (<4 mg dexamethasone/day) for a minimum period of 4 weeks post-treatment are eligible.
12. Pregnant or lactating
13. Treatment with other investigational drugs within 14 days of start of the study drug for non-myelosuppressive agents, and within 28 days of start of the study drug for myelosuppressive agents.
14. Additional criteria for the Combination cohorts: Uncontrolled ascites (defined as 2 or more palliative taps in the last 30 days before screening).
15. Additional criteria for the Combination cohorts with bevacizumab only: uncontrolled clinically significant cardiac disease, hypertension, arrhythmias, or angina pectoris; acute myocardial infarction or cerebrovascular accident within 12 months of initiation of PROMITIL treatment.
16. Additional criteria for the Combination cohorts with bevacizumab only: Any contraindication for treatment with Bevacizumab (e.g active bleeding, recent extensive surgery).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2012-10; Primary Completion 2017-11 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Maximal Tolerated Dose (MTD) of PROMITIL | First cycle of treatment (4 weeks)
  Only DLTs occurring during the first cycle of treatment for each participant will determine MTD endpoint
Dose Limiting Toxicity (DLT) of PROMITIL | First cycle of treatment (4 weeks)
Pharmacokinetic (PK) profile of PROMITIL | 3 cycles of treatment (12 weeks)
  PK assessments will monitor plasma levels of MLP and metabolite (MMC), as well as PK parameters (Cmax, AUC0-t, AUC 0-∞, MRT, t½ , Kel, Cl, VD).

SECONDARY OUTCOMES:
Anti-tumor responses to the delivered PROMITIL regimens | 12 months
Toxicity profile of PROMITIL | 3 cycles of treatment (12 weeks)

CONTACTS AND LOCATIONS:
Locations (4):
- Israel (4):
  - Rambam Health Care Campus, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Chaim Sheba Medical center, Ramat Gan
  - Tel-Aviv Sourasky Medical Center, Tel Aviv

REFERENCES:
- [Derived] Golan T, Grenader T, Ohana P, Amitay Y, Shmeeda H, La-Beck NM, Tahover E, Berger R, Gabizon AA. Pegylated liposomal mitomycin C prodrug enhances tolerance of mitomycin C: a phase 1 study in advanced solid tumor patients. Cancer Med. 2015 Oct;4(10):1472-83. doi: 10.1002/cam4.491. Epub 2015 Jul 14. PMID 26172205